CLINICAL TRIAL: NCT06768073
Title: Clinical Outcomes and Safety of an Intravaginal Negative Pressure Medical Device in the Treatment of Genitourinary Syndrome of Menopause (GSM): A Pilot Study
Brief Title: Intravaginal Negative Pressure Medical Device for Treatment of Genitourinary Syndrome of Menopause (GSM)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AVeta Medical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10510
Record Dates: First submitted 2024-12-13; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Genitourinary Syndrome of Menopause

STUDY DESIGN:
Who Masked: Participant
Masking Description: Randomization with take place after successful screening of the subjects and prior to the first treatment.
  Also, to minimize bias, the clinical exams conducted at the 1-month and 3-month post-treatment visits will be performed by a physician blinded to randomization assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Active Treatment (Experimental): The VITA AV Clinical System (consisting of the VITA AV Probe Kit and the Medela Pump), has a white connector component, part number 10531-01, to allow the vacuum to be delivered to the vaginal tissue when then vacuum pump is activated.
  Interventions: Device: Sham (No Treatment)
- Sham Treatment (Sham Comparator): The VITA AV Clinical System (consisting of the VITA AV Probe Kit and the Medela Pump), has a black connector component, part number 10531-02, to block and prevent the vacuum from being delivered to the vaginal tissue when then vacuum pump is activated.
  Interventions: Device: Sham (No Treatment)

INTERVENTIONS:
Device: Sham (No Treatment) — The Sham device is identified to the Active device with the exception that it has a black connector component, part number 10531-02, to block the vacuum from reaching the vaginal tissue with vacuum pump activation. In this manner, the control procedure has been designed to mimic the active therapy to the extent practicable allowing for subject blinding.

SUMMARY:
This pilot study aims to evaluate the safety and effectiveness of the VITA AV Clinical System over a period of up to three months after the last treatment, compared to a sham device. The study focuses on improving vaginal signs and symptoms of Genitourinary Syndrome of Menopause (GSM) in post-menopausal women who experience moderate to severe pain during intercourse (dyspareunia). Long-term follow-up visits will assess the ongoing effectiveness and durability of the treatment, while also collecting safety data.

DETAILED DESCRIPTION:
There will be up to 6 in-person visits (screening visit, 4 treatment visits and 2 follow-up visits) for all subjects.

Screening After signing the informed consent form, subjects will be screened to ensure they meet the inclusion and exclusion criteria before initiating treatment.

Screening includes collecting information from the patient history (medical history, demographics and medications) as well as conducting the following clinical assessments:

* Dilator suitability.
* Papanicolaou Test (current within last year or repeated within 2 weeks of initial treatment).
* Sexually transmitted infections screening test (gonorrhea, chlamydia, bacterial vaginosis, trichomonas and yeast)
* Pregnancy Test
* Vaginal Health Index (VHI) Score.
* Vaginal pH.
* Clinical examination to confirm that the vaginal canal is free of any lesions other than symptoms of GSM.
* Self-assessment of symptoms related to GSM and confirmation of moderate to severe dyspareunia.

All screening information necessary to evaluate whether the subject meets the inclusion/exclusion criteria should be available and reviewed prior to treatment. Subjects who do not meet the eligibility criteria upon screening will be considered screening failures. Screening failures will not be followed further except in case of adverse events occurring at the screening visit. In this case, subjects will be monitored until the adverse event(s) are resolved.

The eligible subjects will be randomized and introduced to the treatment at the first treatment visit.

Treatment Visits

The following are completed prior to treatment:

1. Pre-Treatment Assessments

   * Urinary Tract Infection Test.
   * Vaginal pH.
   * Vaginal moisture (modified Schirmer Test).
   * Vaginal Maturation Index (VMI) Score.
   * Clinical Examination - Immediately prior to each treatment, a visual examination of the vulvo-vaginal area is carried out. The appearance of the vaginal mucosa before each treatment will be assessed (by the same investigator for each subject) taking parameters of Vaginal Mucosa Assessment (VMA) into account.
   * Vaginal Health Index (VHI) Score.
   * Imaging of Vaginal Wall - An image of the mucosa will be taken after the clinical examination and prior to each treatment.
   * Self-assessment of symptoms related to GSM and confirmation of moderate to severe dyspareunia.
   * Female Sexual Function Index (FSFI) questionnaire.
2. Randomization

Before initiating treatment, subjects continuing to meet eligibility criteria will be randomized to one of following two arms:

* VITA AV Clinical System (active treatment).
* Sham device.

Each active treatment is delivered at a negative pressure of 460 mmHg for 5 minutes. After the treatment, the clinician will re-assess the vaginal mucosa to review the induced micro-trauma, if any. This appears as visible dome shaped effects on the vaginal mucosa corresponding to the apertures in the intravaginal tip. They may appear red indicating induced petechiae, which is the desired response. Images will be taken after each treatment to record the treatment effect at site # 2.

After the initial treatment, each subject returns for an additional 3 treatments performed at 4-week intervals (+/-4 days) for a total of four treatments.

In addition, the following are assessed, as part of the clinical examination, prior to performing subsequent treatments to ensure that the vaginal canal is free from:

1. bleeding,
2. inflammation,
3. the desired microtrauma effects of any previous treatment.
4. other abnormal effects.

Follow-Up Visits:

Will occur at 1-, 3- post the last treatment will take place for all subjects. Will occur at 6-, 9- and 12-months post the last treatment will take place for subjects in the Active treatment only.

Note: The 9-month follow-up visit will be conducted via phone call.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy postmenopausal subjects from 1 to 15 years since their last menstrual cycle.
2. Willingness to refrain from using alternative therapies for treatment of symptoms of GSM, unless medically necessary, through the duration of this study.
3. Moderate to severe dyspareunia associated with GSM. (i.e., ≥4 on the 11-point patient-reported numeric rated dyspareunia scale).
4. Subjects who are sexually active (i.e. have had or have attempted to have sexual activity with vaginal penetration within approximately 1 month of screening visit).
5. Subjects who anticipate engaging or attempting to engage in sexual activity (with vaginal penetration) at least twice a month during the trial.
6. Vaginal Health Index (VHI) score of less than or equal to 15.
7. Vaginal pH >5.0.
8. The subject is anatomically suitable to the intravaginal tip as determined by the Investigator.
9. Normal Papanicolaou test within the past year (or should be done 2 weeks before the trial begins). Subject can ONLY participate on negative results.
10. Vaginal canal free of any lesions other than symptoms of GSM as determined by the Investigator.
11. Negative screening for chlamydia, gonorrhea, bacterial vaginosis, trichomonas and yeast.
12. Willingness and ability to give voluntary written informed consent to participate in the study and comply with protocol requirements.
13. Willingness to refrain from sexual intercourse for at least 48 hours before all visits and for at least 48 hours after all treatments.
14. Willingness to stop using current vaginal lubricant, moisturizers or similar and only use the lubricant provided by the clinic.
15. Willingness to stop using the clinic assigned lubricant for at least 48 hours before all scheduled visits post screening.
16. Willingness to refrain from any pelvic floor therapy for the duration of the trial.
17. Willingness to refrain from enrolling in another clinical trial for the duration of this study.

Exclusion Criteria:

1. Subjects on Hormone Therapies (HT), systemic or local, or within 6 months of cessation of HT prior to inclusion in the study.
2. Subjects with bleeding disorders.
3. Subjects with any sexually transmitted disease.
4. Subjects on prescribed anticoagulants such as antiplatelets and anticoagulants (Heparin, Warfarin, Clopidogrel, Apixaban, Rivaroxaban).
5. Any active genital infections.
6. Abnormal Papanicolaou test within the past year.
7. Positive pregnancy test or planned pregnancy during the study period.
8. Complete procidentia or prolapse that in investigator opinion would be unsuitable for probe placement.
9. Subjects with urogenital sinus (this is when urethral opening is combined with the vagina opening), otherwise the urethral opening will be traumatized potentially resulting in a urinary tract infection (UTI).
10. Subjects with a compromised immune system.
11. Subjects who have undergone pelvic irradiation treatment.
12. Subjects who have undergone off-label procedures such as "vaginal rejuvenation" (e.g., laser or thermoablative techniques).
13. Pelvic surgery within 6 months prior to the start of the study.
14. Undiagnosed vaginal bleeding.
15. Subjects with bleeding during screening examination due to friable vaginal mucosa and/or very thin epithelial layer, such that investigator determines the VITA AV treatment would be contraindicated.
16. Subjects receiving chemotherapy or radiotherapy or subjects with any diagnosed gynecological cancers.
17. History of breast cancer who have had chemotherapy within the last 5 years or are on aromatase inhibitors.
18. Any general health or anatomical conditions, mental health or social situation which, in the opinion of the investigator, could represent an increased risk for the subject, or the ability of the subject to complete study requirements.
19. Currently participating or considering participation in any other research of an investigational drug or device. Does not include observational studies.
20. Subjects that have previously received this treatment as part of a clinical trial.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-03-03 (Estimated); Primary Completion 2025-11-03 (Estimated); Study Completion 2025-11-03 (Estimated)

PRIMARY OUTCOMES:
Safety Evaluation of the VITA AV Clinical System compared to a sham device from baseline to 3-months post the last treatment. | Baseline to 3-months post the last treatment.
  Safety will be assessed by monitoring all adverse events, with particular attention to serious adverse events (SAEs) related to the device or procedure.
Percentage of Vaginal Superficial Cells to evaluate the performance of the VITA AV Clinical System compared to a sham device from baseline to 3-months post the last treatment. | Baseline to 3-months post the last treatment.
  Quantified using cytological analysis to determine the percentage of superficial cells. Changes will be assessed from baseline up to 3 months following the last treatment. To minimize bias, the clinical exams conducted at the 1-month and 3-month post-treatment visits will be performed by a physician blinded to randomization assignment.
Vaginal Moisture Levels to evaluate the performance of the VITA AV Clinical System compared to a sham device from baseline to 3-months post the last treatment. | Baseline to 3-months post the last treatment.
  Measured using the modified Schirmer Test to assess changes in vaginal hydration levels. Changes will be assessed from baseline up to 3 months following the last treatment. To minimize bias, the clinical exams conducted at the 1-month and 3-month post-treatment visits will be performed by a physician blinded to randomization assignment.
Vaginal pH Levels to evaluate the performance of the VITA AV Clinical System compared to a sham device from baseline to 3-months post the last treatment. | Baseline to 3-months post the last treatment.
  Measured by inserting a cotton swab vaginally, and applying it to the vaginal pH strip to determine changes in vaginal acidity. Changes will be assessed from baseline up to 3 months following the last treatment. To minimize bias, the clinical exams conducted at the 1-month and 3-month post-treatment visits will be performed by a physician blinded to randomization assignment.

SECONDARY OUTCOMES:
Vaginal Health Index (VHI) changes from baseline to each visit (treatment phase and up to the 3-month follow-up) for treatment with the VITA AV Clinical System compared to a sham device. | Baseline to 3-months post the last treatment.
  Evaluated using the Vaginal Health Index, which includes assessments of vaginal elasticity, fluid volume, pH, epithelial integrity, and moisture. Changes will be assessed from baseline, at each visit during the treatment phase and up to the 3-month follow-up. To minimize bias, the clinical exams conducted at the 1-month and 3-month post-treatment visits will be performed by a physician blinded to randomization assignment.
Vaginal Maturation Index (VMI) changes from baseline to each visit (treatment phase and up to the 3-month follow-up) for treatment with the VITA AV Clinical System compared to a sham device. | Baseline to 3-months post the last treatment.
  Assessed using cytological analysis to determine the proportion of parabasal, intermediate, and superficial cells. Changes will be assessed from baseline, at each visit during the treatment phase and up to the 3-month follow-up. To minimize bias, the clinical exams conducted at the 1-month and 3-month post-treatment visits will be performed by a physician blinded to randomization assignment.
Vaginal Mucosa Assessment (VMA) changes from baseline to each visit (treatment phase and up to the 3-month follow-up) for treatment with the VITA AV Clinical System compared to a sham device. | Baseline to 3-months post the last treatment.
  Evaluated through clinical examination of the vaginal mucosa, including assessments of atrophy, dryness, and inflammation. Changes will be assessed from baseline, at each visit during the treatment phase and up to the 3-month follow-up. To minimize bias, the clinical exams conducted at the 1-month and 3-month post-treatment visits will be performed by a physician blinded to randomization assignment.
Severity of GSM Symptoms changes from baseline to each visit (treatment phase and up to the 3-month follow-up) for treatment with the VITA AV Clinical System compared to a sham device. | Baseline to 3-months post the last treatment.
  Assessed using a validated symptom severity scale, an 11-point a Visual Analogue Scale (VAS) to evaluate changes in the severity of GSM symptoms.
  Scale breakdown as reported by the subject is as follows: 0 = None (symptom is not present); 1 - 3 = Mild; 4 - 6 = Moderate; and 7 - 10 = Severe.
  Changes will be assessed from baseline, at each visit during the treatment phase and up to the 3-month follow-up.
Durability of Benefit from baseline to each visit (treatment phase and up to the 3-month follow-up) for treatment with the VITA AV Clinical System compared to a sham device. | Baseline to 3-months post the last treatment.
  Assessed using a subject-completed questionnaire to determine the perceived benefit from the treatment and the duration of its effects. Changes will be assessed from baseline, at each visit during the treatment phase and up to the 3-month follow-up.
Female Sexual Function Index (FSFI) from baseline to each visit (treatment phase and up to the 3-month follow-up) for treatment with the VITA AV Clinical System compared to a sham device. | Baseline to 3-months post the last treatment.
  Assessed using the FSFI to evaluate changes in sexual function, including domains such as desire, arousal, lubrication, orgasm, satisfaction, and pain. Changes will be assessed from baseline, at each visit during the treatment phase and up to the 3-month follow-up.

OTHER OUTCOMES:
Long-term Safety Evaluation of the VITA AV Clinical System Treatment. | Baseline to 12-months post the last treatment
  Safety will be assessed by monitoring all adverse events, with particular attention to serious adverse events (SAEs) related to the device or procedure.
Percentage of Vaginal Superficial Cells to evaluate the Long-term Clinical Efficacy of the VITA AV Clinical System Treatment. | Baseline to 12-months post the last treatment.
  Quantified using cytological analysis to determine the percentage of superficial cells.
Vaginal Moisture Levels to evaluate the Long-term Clinical Efficacy of the VITA AV Clinical System Treatment. | Baseline to 12-months post the last treatment.
  Measured using the modified Schirmer Test to assess changes in vaginal hydration levels.
Vaginal pH Levels to evaluate the the Long-term Clinical Efficacy of the VITA AV Clinical System Treatment. | Baseline to 12-months post the last treatment.
  Measured by inserting a cotton swab vaginally, and applying it to the vaginal pH strip to determine changes in vaginal acidity.
Vaginal Health Index (VHI) changes to evaluate the the Long-term Clinical Efficacy of the VITA AV Clinical System Treatment. | Baseline to 12-months post the last treatment.
  Evaluated using the Vaginal Health Index, which includes assessments of vaginal elasticity, fluid volume, pH, epithelial integrity, and moisture.
Vaginal Maturation Index (VMI) changes to evaluate the the Long-term Clinical Efficacy of the VITA AV Clinical System Treatment. | Baseline to 12-months post the last treatment.
  Assessed using cytological analysis to determine the proportion of parabasal, intermediate, and superficial cells.
Vaginal Mucosa Assessment (VMA) changes to evaluate the the Long-term Clinical Efficacy of the VITA AV Clinical System Treatment. | Baseline to 12-months post the last treatment.
  Evaluated through clinical examination of the vaginal mucosa, including assessments of atrophy, dryness, and inflammation.
Severity of GSM Symptoms changes to evaluate the the Long-term Clinical Efficacy of the VITA AV Clinical System Treatment. | Baseline to 12-months post the last treatment.
  Assessed using a validated symptom severity scale, an 11-point a Visual Analogue Scale (VAS) to evaluate changes in the severity of GSM symptoms.
  Scale breakdown as reported by the subject is as follows: 0 = None (symptom is not present); 1 - 3 = Mild; 4 - 6 = Moderate; and 7 - 10 = Severe.
Female Sexual Function Index (FSFI) to evaluate the Long-term Clinical Efficacy of the VITA AV Clinical System Treatment. | Baseline to 12-months post the last treatment.
  Assessed using the FSFI to evaluate changes in sexual function, including domains such as desire, arousal, lubrication, orgasm, satisfaction, and pain.
Long-term Durability of Benefit of the VITA AV Clinical System Treatment. | Baseline to 12-months post the last treatment.
  Assessed using a subject-completed questionnaire to determine the perceived benefit from the treatment and the duration of its effects.
Subject Satisfaction | 6-month to 12-month follow-up visits
  Assessed using a subject-completed questionnaire for Active Arm of study to determine the perceived level of satisfaction of the VITA AV Clinical System Treatment using the following 5 ratings: Poor; Fair; Good; Very good and Excellent.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Philips, Principal Investigator — IMA Clinical Research
Locations (2):
- IMA Clinical Research,, Warren Township, New Jersey, United States
- Pineo Clinic (Pineo Medical Ecosystem), Tbilisi, Georgia